CLINICAL TRIAL: NCT01354613
Title: Reduced Contractile Reserve: a Therapeutic Target in Heart Failure With Preserved Ejection Fraction
Brief Title: Reduced Contractile Reserve: a Therapeutic Target in Heart Failure With Preserved Ejection Fraction(HFpEF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-2010-0061; R21HL106103-01 (NIH)
Record Dates: First submitted 2011-05-05; First posted 2011-05-17 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Pulmonary Disease; Left Ventricular Hypertrophy/Hypertension
MeSH Terms: conditions — Lung Diseases; Hypertrophy, Left Ventricular; Hypertension | interventions — Dobutamine; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HFpEF (Experimental): 25 patients with clinically diagnosed heart failure with preserved ejection fraction, confirmed by Framingham criteria, with EF > 50% and without evidence of active ischemia or known severe CAD, valvular or pericardial disease, infiltrative or hypertrophic cardiomyopathy, cor pulmonale, severe pulmonary disease, or primary renal disease. Subjects will receive amlodipine, oral administration for a period of 12 weeks.
  Interventions: Drug: Dobutamine; Drug: Amlodipine
- Pulmonary Disease (Experimental): 20 patients with pulmonary disease and no clinical evidence of cardiovascular disease
  Interventions: Drug: Dobutamine
- LVH/HTN (Experimental): 20 subjects with known left ventricular hypertrophy and clinically diagnosed hypertension without the diagnosis of heart failure.
  Interventions: Drug: Dobutamine
- HFpEF placebo (Placebo Comparator): 25 patients with clinically diagnosed heart failure with preserved ejection fraction, confirmed by Framingham criteria, with EF > 50% and without evidence of active ischemia or known severe CAD, valvular or pericardial disease, infiltrative or hypertrophic cardiomyopathy, cor pulmonale, severe pulmonary disease, or primary renal disease. Subjects will be administered a placebo for a period of 12 weeks.
  Interventions: Drug: Dobutamine

INTERVENTIONS:
Drug: Dobutamine — IV administration at the initial study visit (all groups) and at the final study visit for the drug intervention arm (HFpEF group only). Administration of low-dose dobutamine at 5mcg/kg/min and 10mcg/kg/min for periods of approximately 30minutes/dose for purposes of performing a low-dose stress exam on the heart.
Drug: Amlodipine — Participants will be randomized to treatment with either amlodipine 5 mg daily or placebo, in double-blind fashion, 25 patients in each group. 12 week oral administration of 5mg/day, uptitrated to 10mg/day, determined by PI.
  Arms: HFpEF

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) accounts for over 50% of heart failure cases in the United States, affecting a primarily elderly population. No treatment has been shown to affect mortality in HFpEF, which is more than 50% at five years a hospitalization. This project explores the underlying cardiovascular physiology of patients with HFpEF with the goal of identifying new therapeutic targets that would allow improved treatment of this devastating disease.

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction (HFpEF) is a difficult disease to diagnose due to nonspecific symptoms and clinical findings. The disease occurs in the elderly, who often have other illnesses and signs of aging that make diagnosis of heart failure more difficult. Recently, it has been suggested that HFpEF, which has primarily been thought to be a diastolic disease, is in fact multifactorial, with elements of abnormal systolic function and increased vascular stiffness playing a role in disease pathology. No treatment has been shown to reduce the high mortality of the disease. However, few studies have evaluated this population of patients during periods of increased physiologic stress, despite the consistent clinical presentation of impaired exercise tolerance with few symptoms at rest. This study explores the multifactorial physiology of HFpEF, with a detailed investigation of the specificity of abnormalities in contractile reserve and vascular stiffness for this disease, and exploration of the modifiability of these abnormalities. The techniques used are non-invasive, involving echocardiographic evaluation of cardiac function, and measurement of arterial stiffness using tonometry. The first aim of the study is to explore the specificity of a potential diagnostic test for HFpEF by investigating the change in ejection fraction before and after β-adrenergic stimulation with low-dose dobutamine in HFpEF compared to other groups important to distinguish clinically, specifically patients with shortness of breath due to pulmonary disease, and those with hypertension and left ventricular hypertrophy without clinical heart failure. In the second aim, the study will investigate the ability of the calcium channel blocker, amlodipine, to restore normal contractile responses of the myocardium. In the third aim, the role of arterial stiffness in drug responses in HFpEF will be explored. It is anticipated that improved understanding of the complex physiology of this multifactorial disease gained through this study will lead to more rational design of large clinical trials studying promising agents for HFpEF that impact not only diastolic function, but contractile reserve and arterial properties as well.

ELIGIBILITY:
Inclusion Criteria:

* Male or female; Age 18 or older.
* Left ventricular ejection fraction ≥ 50%.
* Symptomatic heart failure or appropriate comparator group criteria
* Informed consent signed by the subject

Exclusion Criteria:

* Symptoms of active ischemia.
* Moderate or severe mitral or aortic stenosis, or severe aortic insufficiency.
* Serum creatinine > 3.0 or chronic hemodialysis.
* Known chronic hepatic disease; defined as aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels > 3.0 times the upper limit of normal as read at the local lab.
* Severe renal dysfunction, i.e. glomerular filtration rate (GFR) <30 ml/min.
* Atrial fibrillation
* Myocardial infarction within the last year
* Coronary bypass surgery within the last 6 months
* Stroke within the last 6 months
* Known aortic aneurysm
* Contra-indication to withdrawal of beta blocker or antihypertensive medications
* Resting or orthostatic hypotension (SBP < 90 mmHg)
* Any gastrointestinal disorder which would interfere with drug absorption
* Any significant valvular heart disease, including prior multiple valve replacement.
* Pericardial Disease
* Infiltrative or hypertrophic cardiomyopathy
* Cor pulmonale
* Unstable coronary disease
* Pregnancy
* Any condition which may prevent the subject from adhering to the study protocol, as determined by the investigator

Heart Failure with Preserved Ejection Fraction

* Clinical evidence of heart failure with preserved ejection fraction, as manifest by at least 2 symptoms or signs, including dyspnea on exertion or at rest, orthopnea, jugular venous distention or hepatojugular reflux, rales or edema.
* Controlled systolic BP (< 150 mmHg on the day of study)

Pulmonary Disease Group

* Known obstructive airways disease with objective documentation of an isolated obstructive defect by pulmonary function testing.
* No history of heart failure.
* No history of cardiovascular disease, with the exception of hypertension or hyperlipidemia
* History and physical examination free of signs and symptoms of heart failure, including elevated jugular venous pressure, hepatojugular reflux, rales or edema.
* Baseline echocardiographic examination without evidence of heart failure, including systolic dysfunction of the LV or RV, or evidence of more than mild diastolic dysfunction on non-invasive assessment.

HTN/LVH Group

* Known history of hypertension.
* Echocardiographic evidence of left ventricular hypertrophy and diastolic dysfunction.
* No history or physical examination evidence of heart failure, including excessive dyspnea on exertion, dyspnea at rest, orthopnea, PND, jugular venous distention, hepatojugular reflux, rales or edema.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in ejection fraction with 5mcg/kg/min dobutamine | day 0 and 12 week study visit
  The primary outcome variable in this analysis will be change in ejection fraction from baseline at the 5 mcg dobutamine dose.
Change in pulse wave velocity | 12 week study visit
  Change in carotid-femoral pulse wave velocity (PWV) with 12 weeks of therapy with amlodipine or placebo will be the primary outcome variable.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy K Sweitzer, MD, PhD, Principal Investigator — UW-Madison
Locations (1):
- UW - Madison, Madison, Wisconsin, United States